CLINICAL TRIAL: NCT00582894
Title: Reduced-Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Malignant Hematological Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: George Selby, MD, University of Oklahoma Health Sciences Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Reduced-Intensity; IRB #11835 (Other: University of Oklahoma Health Sciences Center)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Hematological Neoplasms; Hematopoietic Stem Cell Transplantation
Keywords: Allogenic stem cell transplant; Hematologic diseases
MeSH Terms: conditions — Hematologic Neoplasms; Hematologic Diseases | interventions — Busulfan; fludarabine; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other): Preparative regimen of 1)Busulfex 3.2 mg/kg/day for 2 days, infused over 3 hours, on Day-6 and Day-5 2)Fludarabine 30 mg/m2/day for 5 days on Day-6 to D-2 and 3) Alemtuzumab 10 mg/day IV on days - 5 to -1
  Interventions: Drug: Busulfex, Fludarabine, ALemtuzumab

INTERVENTIONS:
Drug: Busulfex, Fludarabine, ALemtuzumab — Busulfex 3.2 mg/kg/day for 2 days infused over 3 hours, Days -6 and Day-5 Fludarabine 30 mg/m2/day for 5 days on Day -6 to D-2 Alemtuzumab 10 mg/day IV on Days -5 to -1

SUMMARY:
To evaluate engraftment and toxicity of a reduced intensity preparative regimen for patients who receive a matched related or unrelated donor allogeneic stem cell transplant (ASCT) for malignant hematological diseases

DETAILED DESCRIPTION:
Primary Endpoints:

1. Engraftment of donor cells
2. Regimen related toxicities

Secondary Endpoints:

1. Disease-free survival
2. Overall survival

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0-2
* Ejection fraction > 30%
* AST/ALT and bilirubin not > 4 times normal
* Creatinine clearance greater than 70 ml/min.
* FEV1 greater than 1.0 and diffusion capacity greater than 40%
* Age 18-75 years
* Patients must be at high risk for conventional regimen related toxicity
* Malignant hematologic disease that would otherwise be considered treatable with ASCT

Exclusion Criteria:

* Does not meet the above Inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Selby, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began February 2005 and concluded around March 2007
Groups:
- Reduced Intensity Regimen: Preparative regimen of 1)Busulfex 3.2 mg/kg/day for 2 days, infused over 3 hours, on Day-6 and Day-5 2)Fludarabine 30 mg/m2/day for 5 days on Day-6 to D-2 and 3) Alemtuzumab 10 mg/day IV on days - 5 to -1
Period: Overall Study
Arm/Group | Reduced Intensity Regimen
Started | 17
Day 100 Post Transplant | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Transplant Related Mortality (TRM)
Time Frame: At Day 100 post trans-plant
Measure: Number; unit: Participants
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Number of Participants Relapse-Free
Time Frame: 100 days post-transplant
Population: Last observation carried forward
Measure: Number; unit: Participants
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 17
Participants | 5

3. Primary Outcome: Number of Participants Experiencing Engraftment Donor Chimerism (EDC)
Time Frame: At time of study termination
Measure: Number; unit: Participants
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 17
Participants | 17

4. Secondary Outcome: Number of Participants Overall Survival as a Function of Time.
Time Frame: 100 days post transplant
Population: Last observation carried forward
Measure: Number; unit: Participants
Arm/Group | Reduced Intensity Regimen
Number analyzed (Participants) | 17
Participants | 11

ADVERSE EVENTS:
Time Frame: Day 100 Post Transplant
Arm/Group | Reduced Intensity Regimen
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Regimen (N=17)
Intracranial hemorrhage - recurrence (Vascular disorders) | 1 (1) — Event determined to be "not related" to study participation; resulted in death of participant
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Regimen (N=17)
Positive Cytomegalovirus cultures (Blood and lymphatic system disorders) | 1 (1) — Hospitalized for treatment and recovered without sequelae
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Hospitalized and recovered without sequelae
Blasts in bone marrow (Blood and lymphatic system disorders) | 1 (1) — Determined to be not related to study participation; recovered without sequelae
Syncopal episode / Hypotension (General disorders) | 1 (1) — Determined to be "not related" to study participation; recovered without sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes